CLINICAL TRIAL: NCT01627691
Title: REPRISE II: REpositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of Lotus™ Valve System - Evaluation of Safety and Performance
Brief Title: REPRISE II: REpositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of Lotus™ Valve System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP3687; TP3687 (Other: Boston Scientific)
Record Dates: First submitted 2012-06-05; First posted 2012-06-26 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lotus Valve System (Experimental): Patients enrolled will receive the Lotus Valve.
  Interventions: Device: Lotus Valve System

INTERVENTIONS:
Device: Lotus Valve System — * bioprosthetic bovine pericardial aortic valve
  * delivery system

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Lotus™ Valve System for transcatheter aortic valve replacement (TAVR) in symptomatic subjects with severe calcific aortic stenosis who are considered high risk for surgical valve replacement.

DETAILED DESCRIPTION:
The REPRISE II clinical study is a prospective, single-arm, multicenter study designed to evaluate the safety and performance of the Lotus Valve System for TAVR in symptomatic subjects who have severe calcific aortic valve stenosis and who are at high risk for surgical aortic valve replacement (SAVR).

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥70 years of age
* Subject has documented calcific native aortic valve stenosis
* Subject has a documented aortic annulus size between ≥19 and ≤27 mm based on pre-procedure diagnostic imaging
* Symptomatic aortic valve stenosis with NYHA Functional Class ≥ II
* Subject is considered high risk for surgical valve replacement
* Heart team assessment that the subject is likely to benefit from valve replacement.
* Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
* Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

* Subject has a congenital unicuspid or bicuspid aortic valve.
* Subject with an acute myocardial infarction within 30 days of the index procedure
* Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months, or has any permanent neurologic defect prior to study enrollment.
* Subject is on dialysis or has serum creatinine level >3.0 mg/dL or 265 µmol/L.
* Subject has a pre-existing prosthetic heart valve (aortic or mitral) or a prosthetic ring in any position.
* subject cannot have more than moderate mitral, aortic or tricuspid regurgitation
* Subject has a need for emergency surgery for any reason.
* Subject has a history of endocarditis within 12 months of index procedure or evidence of an active systemic infection or sepsis.
* Subject has echocardiographic evidence of intra-cardiac mass, thrombus or vegetation.
* Subject has low Hgb, platelet count or >700,000 cells/mm3, or low white blood cell count.
* Subject requires chronic anticoagulation therapy and cannot tolerate concomitant therapy with either aspirin or clopidogrel/ticlopidine
* Subject has active peptic ulcer disease or gastrointestinal bleed within the past 3 months, other bleeding diathesis or coagulopathy or will refuse transfusions.
* Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all thienopyridines, heparin, nickel, tantalum, titanium, or polyurethanes.
* Subject has a life expectancy of less than 12 months due to non-cardiac, co-morbid conditions based on the assessment of the investigator at the time of enrollment.
* Subject has hypertrophic obstructive cardiomyopathy.
* Subject has any therapeutic invasive cardiac procedure within 30 days prior to the index procedure (except for pacemaker implantation which is allowed).
* Subject has untreated coronary artery disease.
* Subject has documented left ventricular ejection fraction <30%.
* Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
* Subject has severe peripheral vascular disease or symptomatic carotid or vertebral disease.
* Narrow Femoral artery lumen precludes the use of either Lotus device size, or severe iliofemoral tortuosity or calcification that would prevent safe placement of the introducer sheath.
* Current problems with substance abuse (e.g., alcohol, etc.).
* Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
* Patient has preexisting untreated conduction system disorder that requires new pacemaker implantation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-10-08 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Dumonteil, MD, Principal Investigator — Clinique Pasteur
Locations (20):
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Brisbane
  - Monash Medical Center, Melbourne
  - St. Vincent's Hospital, Melbourne
- France (5):
  - Hôpital Cardiologique CHRU de Lille, Lille
  - Hôpital Cardiologique de Lyon, Lyon
  - Institut Cardiovasculaire Paris Sud, Paris
  - Centre Hôpital Universitaire Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (2):
  - Deutsches Herzzentrum München, München
  - Helios Klinikum Siegburg, Siegburg
- Ospedale Ferrarotto, Catania, Italy
- Erasmus MC - Thorax Center, Rotterdam, Netherlands
- Hospital Clinico San Carlos, Madrid, Spain
- University Hospital of Lund, Lund, Sweden
- INSELSPITAL - Universitätsspital Bern, Bern, Switzerland
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - Royal Sussex County Hospital, Brighton
  - The General Infirmary, Leeds
  - Guys and St. Thomas NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meredith IT, Walters DL, Dumonteil N, Worthley SG, Tchetche D, Manoharan G, Blackman DJ, Rioufol G, Hildick-Smith D, Whitbourn RJ, Lefevre T, Lange R, Muller R, Redwood S, Feldman TE, Allocco DJ, Dawkins KD. 1-Year Outcomes With the Fully Repositionable and Retrievable Lotus Transcatheter Aortic Replacement Valve in 120 High-Risk Surgical Patients With Severe Aortic Stenosis: Results of the REPRISE II Study. JACC Cardiovasc Interv. 2016 Feb 22;9(4):376-384. doi: 10.1016/j.jcin.2015.10.024. PMID 26892084
- [Derived] Meredith Am IT, Walters DL, Dumonteil N, Worthley SG, Tchetche D, Manoharan G, Blackman DJ, Rioufol G, Hildick-Smith D, Whitbourn RJ, Lefevre T, Lange R, Muller R, Redwood S, Allocco DJ, Dawkins KD. Transcatheter aortic valve replacement for severe symptomatic aortic stenosis using a repositionable valve system: 30-day primary endpoint results from the REPRISE II study. J Am Coll Cardiol. 2014 Sep 30;64(13):1339-48. doi: 10.1016/j.jacc.2014.05.067. PMID 25257635

RESULTS

PARTICIPANT FLOW:
Groups:
- REPRISE II and Extension Overall: Transcatheter aortic valve replacement (TAVR) with the Lotus™ Valve System.
  Lotus Valve System: - bioprosthetic bovine pericardial aortic valve
  - delivery system
Period: Overall Study
Arm/Group | REPRISE II and Extension Overall
Started | 250
Primary Endpoint (30days) | 239
Completed | 232
Not Completed | 18
Not completed — Death | 11
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Missed the visit | 3

BASELINE CHARACTERISTICS:
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Unknown or not reported | 250
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 74
  Europe | 171
EuroSCORE [Mean (Standard Deviation); unit: percent predicted mortality] — The European System for Cardiac Operative Risk Evaluation is a risk model where if a risk factor is present in a subject, a weight or number is assigned. The weights are added to give an approximate percent predicted mortality. A higher score means a higher risk and a lower score means a lower risk.
  percent predicted mortality | 6.4 (6.2)
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons Score is a risk model used to predict a subject's risk of mortality and morbidities for the most commonly performed cardiac surgeries. The model is a percentage score from 0 to 100 where a lower score means a lower risk and higher score means a higher risk."
  units on a scale | 6.5 (4.2)
NYHA Functional Class [Count of Participants; unit: Participants] — New York Heart Association Classification is a system for defining cardiac disease and related functional limitations into four broad categorizations. The categories range from NYHA I (No limitations) to NYHA IV (inability to carry out any physical activity without discomfort).
  Participants
    Grade I | 0
    Grade II | 57
    Grade III | 166
    Grade IV | 27

OUTCOME MEASURES:

1. Primary Outcome: Primary Device Performance Endpoint: Mean Aortic Valve Pressure Gradient at 30 Days Post Implant Procedure
Description: Mean aortic valve pressure gradient at 30 days post implant procedure as measured by echocardiography and assessed by an independent core laboratory.
Time Frame: 30 days
Population: As specified, this endpoint was evaluated using data from the first 120 patients enrolled in the study
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 120
mmHG | 11.45 (5.20)

2. Primary Outcome: Primary Safety Endpoint: All-cause Mortality at 30 Days Post Implant Procedure
Description: Mortality at 30 days from all patients enrolled in the study (ITT population): the proportion of patients who experience an event through 30 days post-procedure out of the patients who have either had an event within 30 days post-procedure or who were event-free with last follow-up at least 23 days post-procedure
Time Frame: 30 days
Population: Mortality at 30 days from all patients enrolled in the study (ITT population): the proportion of patients who experience an event through 30 days post-procedure out of the patients who have either had an event within 30 days post-procedure or who were event-free with last follow-up at least 23 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 249
Participants | 11

3. Secondary Outcome: Effective Orifice Area
Description: Effective orifice area measured by echocardiography at 30 days and assessed by an independent core laboratory (ITT population)
Time Frame: 30 days
Population: Patients with an echocardiography available from the 30-day follow-up visit and analyzable by the Core Lab
Measure: Mean (95% Confidence Interval); unit: square centimeter
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 170
square centimeter | 1.73 [1.66 to 1.79]

4. Secondary Outcome: Device Performance Endpoint: Successful Vascular Access
Description: Successful vascular access, delivery and deployment of the Lotus Valve System and successful retrieval of the delivery system as reported from site
Time Frame: Post-procedure
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 250
Participants | 247

5. Secondary Outcome: Device Performance Endpoint: Successful Retrieval
Description: Successful retrieval (complete resheathing of the Lotus valve in the catheter and removal from the body) of the Lotus Valve System if retrieval is attempted, as reported from site
Time Frame: Post-procedure
Population: Number of participants for whom a retrieval of the valve was attempted
Measure: Count of Participants; unit: Participants
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 13
Participants | 12

6. Secondary Outcome: Device Performance Endpoint: Successful Repositioning
Description: Successful repositioning (partial or complete resheathing of the Lotus Valve in the catheter and redeployment in a more accurate position within the aortic valve annulus) of the Lotus Valve System if repositioning is attempted for the last valve attempted, as reported from site
Time Frame: Post-procedure
Population: Number of participants for whom a repositioning of the valve was attempted
Measure: Count of Participants; unit: Participants
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 85
Participants | 85

7. Secondary Outcome: Device Success According to the Valve Academic Research Consortium (VARC)
Description: Absence of procedural mortality as reported from site AND Correct positioning of a single prosthetic heart valve into the proper anatomical location as reported from site AND Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation as measured from an independent core lab on the post-procedure echocardiography)
Time Frame: Post-procedure
Population: Number of patients who had an echocardiography available post-procedure for the Core Lab to measure the performance of the prosthetic heart valve as described above
Measure: Count of Participants; unit: Participants
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 175
Participants | 96

8. Secondary Outcome: Grade of Aortic Valve Regurgitation
Description: Grade of paravalvular aortic valve regurgitation at 30 days as measured by echocardiography and assessed by an independent core laboratory
Time Frame: 30 days
Population: Patients with echocardiography available from the 30-day follow-up visit and analyzable from the Core Lab for those measurements
Measure: Count of Participants; unit: Participants
Arm/Group | REPRISE II and Extension Overall
Number analyzed (Participants) | 210
Participants
  None | 159
  Trace/Trivial | 18
  Mild | 31
  Mild-moderate | 0
  Moderate | 1
  Moderate-Severe | 0
  Severe | 0
  Severity not evaluable | 1

ADVERSE EVENTS:
Time Frame: Primary Endpoint (30days)
Arm/Group | REPRISE II and Extension Overall
All-Cause Mortality (participants affected / at risk) | 11/250
Serious Adverse Events (participants affected / at risk) | 152/250
Other Adverse Events (participants affected / at risk) | 157/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REPRISE II and Extension Overall (N=250)
Total (Cardiac disorders) | 97 (123)
Atrioventricular block complete (Cardiac disorders) | 47 (47)
Atrial fibrillation (Cardiac disorders) | 7 (7)
Bundle branch block left (Cardiac disorders) | 7 (7)
Atrioventricular block (Cardiac disorders) | 6 (6)
Cardiac tamponade (Cardiac disorders) | 6 (6)
Cardiac arrest (Cardiac disorders) | 5 (5)
Atrioventricular block first degree (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 2 (2)
Left ventricular failure (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac perforation (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Coronary ostial stenosis (Cardiac disorders) | 1 (1)
Electromechanical dissociation (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Trifascicular block (Cardiac disorders) | 1 (1)
Ventricle rupture (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Total (General disorders) | 26 (28)
Catheter site haematoma (General disorders) | 12 (12)
Catheter site haemorrhage (General disorders) | 7 (7)
Pyrexia (General disorders) | 3 (3)
Puncture site haemorrhage (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Implant site discharge (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Total (Vascular disorders) | 27 (27)
Haemorrhage (Vascular disorders) | 6 (6)
Hypotension (Vascular disorders) | 6 (6)
Femoral artery dissection (Vascular disorders) | 5 (5)
Haematoma (Vascular disorders) | 3 (3)
Angiopathy (Vascular disorders) | 2 (2)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Total (Nervous system disorders) | 16 (19)
Cerebrovascular accident (Nervous system disorders) | 6 (6)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Cerebellar haematoma (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Motor neurone disease (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Total (Infections and infestations) | 18 (18)
Pneumonia (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Bronchiectasis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Puncture site infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Total (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Total (Blood and lymphatic system disorders) | 12 (12)
Anaemia (Blood and lymphatic system disorders) | 8 (8)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 (4)
Total (Injury, poisoning and procedural complications) | 9 (9)
Device failure (Injury, poisoning and procedural complications) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 (1)
Device migration (Injury, poisoning and procedural complications) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Total (Gastrointestinal disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Intestinal functional disorder (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Total (Investigations) | 8 (8)
Haemoglobin decreased (Investigations) | 6 (6)
C-reactive protein increased (Investigations) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1)
Total (Psychiatric disorders) | 5 (5)
Delirium (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Total (Renal and urinary disorders) | 4 (4)
Bladder disorder (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Total (Eye disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1)
Total (Congenital, familial and genetic disorders) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1)
Total (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Total (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Total (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Total (Reproductive system and breast disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Total (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REPRISE II and Extension Overall (N=250)
Total (Cardiac disorders) | 106 (129)
Bundle branch block left (Cardiac disorders) | 98 (99)
Atrioventricular block first degree (Cardiac disorders) | 17 (17)
Atrial fibrillation (Cardiac disorders) | 13 (13)
Total (General disorders) | 61 (98)
Catheter site haematoma (General disorders) | 35 (48)
Catheter site haemorrhage (General disorders) | 25 (26)
Pyrexia (General disorders) | 23 (24)
Total (Vascular disorders) | 35 (35)
Hypertension (Vascular disorders) | 18 (18)
Hypotension (Vascular disorders) | 17 (17)
Total (Infections and infestations) | 19 (19)
Urinary tract infection (Infections and infestations) | 19 (19)
Total (Blood and lymphatic system disorders) | 17 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT01627691/Prot_SAP_000.pdf